CLINICAL TRIAL: NCT03699514
Title: Post Hoc Analysis and Clinical Data Collection for Subjects Tested With Brain Network Activation (BNA™) Technology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ElMindA Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ELM-52
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Healthy; Cognitive Impairment; Neurological Disorder
Keywords: Brain Network Activation (BNA™); EEG; Cognitive Tasks
MeSH Terms: conditions — Cognitive Dysfunction; Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subject who completed or will complete a BNA test
  Interventions: Device: Brain Network Activation (BNA™) technology

INTERVENTIONS:
Device: Brain Network Activation (BNA™) technology — The BNA™ technology was developed and is utilized by ElMindA Ltd. The BNA Analysis System is cleared for use by qualified medical professionals for the post hoc statistical analysis of the human electroencephalogram ("EEG"), utilizing evoked response potentials ("ERP'). This device is indicated for use in individuals 14 to 24 years of age. The BNA Analysis System is to be used with the auditory oddball task only.

SUMMARY:
The study is designed to collect data that will aid in future scientific and engineering exploration of correlations between clinical assessments and BNA scores. The results are primarily intended for scientific inquiry and engineering development purposes, and may be used in future regulatory submissions.

DETAILED DESCRIPTION:
A multi-center study in which subjects that had completed or are completing a BNA test with the Auditory Oddball task (or other tests that will be commercially cleared at any given time), will have the option to complete additional investigational tasks and optional clinical assessments and questionnaire forms. At each site, these additional assessments will be suggested by the site's study doctor or clinician and will be collected with the site's ePRO device. The study will include up to 10,000 subjects which had completed or will complete a standard BNA test. Authorized personnel will offer the subjects to participate in the study immediately after testing or contacting subjects that had completed the test in the past. Procedure of consent will be performed by the PI or delegates.

ELIGIBILITY:
Inclusion Criteria:

* Completed or will complete a BNA test
* Able to speak, read and understand English sufficiently to understand the nature of the study, and to allow completion of all study assessments.
* Willingness to participate

Exclusion Criteria:

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who completed or will complete a BNA test with the Auditory Oddball Task, from both genders, aged 8-99 years.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Engineering development according to clinical assessments | 5 years
  The study is designed to collect data that will aid in future scientific and engineering exploration of correlations between clinical assessments and BNA scores. The results are primarily intended for scientific inquiry and engineering development purposes, and may be used in future regulatory submissions.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Kadima Neuopsychiatry Institute, La Jolla, California
  - Collaborative Behavioral Health, LLC, Chicago, Illinois
  - Collaborative Behavioral Health, LLC, Skokie, Illinois
  - Alivation Health, LLC, Lincoln, Nebraska